CLINICAL TRIAL: NCT02769689
Title: Once a Month High-dose Methylprednisolone During Wash-out Period Between Natalizumab and Fingolimod Treatments in Patients With Multiple Sclerosis: a Randomised, Controlled, Double-blind Trial (NTZ2FTY)
Brief Title: Methylprednisolone During the Switch Between Natalizumab and Fingolimod
Acronym: NTZ2TTY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0259; 2015-003298-14 (Registry Identifier: 2015-003298-14)
Record Dates: First submitted 2016-03-17; First posted 2016-05-12 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Natalizumab; Fingolimod; Methylprednisolone
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylprednisolone; Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Experimental): The primary purpose of this protocol is to investigate the impact of high dose of oral methylprednisolone, given once a month during the washout period between NTZ and Fingolimod (FTY).
  Interventions: Drug: Methylprednisolone; Drug: natalizumab (NTZ); Drug: fingolimob (FTY)
- Placebo (Placebo Comparator): Included patients will receive either methylprednisolone (1 gramme, 1 day every 4 weeks for a total of 3 grammes) or undistinguishable capsules of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Included patients will receive either methylprednisolone (1 gramme, 1 day every 4 weeks for a total of 3 grammes) or undistinguishable capsules of placebo
  Arms: Methylprednisolone
Drug: Placebo — Included patients will receive either methylprednisolone (1 gramme, 1 day every 4 weeks for a total of 3 grammes) or undistinguishable capsules of placebo
  Arms: Placebo
Drug: natalizumab (NTZ) — Patients with MS receiving NTZ for at least 18 months and without any disease activity during the previous year will be eligible. Included patients will receive either methylprednisolone (1 gramme, 1 day every 4 weeks for a total of 3 grammes) or undistinguishable capsules of placebo
  Arms: Methylprednisolone
Drug: fingolimob (FTY) — Every patient will initiate a treatment with FTY 7 weeks after the last NTZ perfusion. Methylprednisolone or placebo will be taken 4, 8 and 12 weeks (W4, W8 and W12) after NTZ discontinuation.
  Arms: Methylprednisolone

SUMMARY:
Progressive multifocal leukoencephalopathy (PML) is the most feared complication when natalizumab (NTZ) is used in the treatment of relapsing multiple sclerosis (MS). The risk of PML increases after 18 months of treatment. When switching from NTZ to another disease modifying treatment (DMT) in these MS patients with an active disease, there is a high risk of inflammatory reactivation. Nonetheless, a washout period of several weeks is necessary before initiating a new DMT.

The primary purpose of this protocol is to investigate the impact of high dose of oral methylprednisolone, given once a month during the washout period between NTZ and Fingolimod (FTY).

DETAILED DESCRIPTION:
Patients with MS receiving NTZ for at least 18 months and without any disease activity during the previous year will be eligible. Included patients will receive either methylprednisolone (1 gramme, 1 day every 4 weeks for a total of 3 grammes) or undistinguishable capsules of placebo.

Every patient will initiate a treatment with FTY 7 weeks after the last NTZ perfusion. Methylprednisolone or placebo will be taken 4, 8 and 12 weeks (W4, W8 and W12) after NTZ discontinuation.

A spinal and brain MRI will be performed at baseline (last NTZ perfusion, noted W0) and 16 to 18 weeks after. The last clinical follow-up will be made after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-Remitting Multiple Sclerosis (Mc Donald's 2010 criteria)
* EDSS<6.0
* At least18 natalizumab infusions
* Planned switch from natalizumab to fingolimod
* Aged between 18 and 65
* Patients must have received high dose IV methylprednisolone during the 5 previous years

Exclusion Criteria:

* Progressive MS
* Uncontrolled MS with natalizumab (existence of a relapse during the previous 12 months or existence of a gadolinium enhancing lesion on a MRI performed during the last 12 months)
* SEP de forme progressive
* Contra-indication to the use of high dose oral methylprednisolone
* Marked cognitive impairment altering protocole understanding
* Switch from natalizumab to a disease modifying treatment different from fingolimod
* Contra-indication to fingolimod use
* Existence of a disease or condition that could alter study completion
* Chronic treatment with steroids
* Acute treatment with steroids (more than 300mg during the month prior to inclusion)
* Contra-indication to gadolinium containing products injection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
efficacy of high dose methylprednisolone compared to that of a placebo | at 6 months
  To evaluate the efficacy of high dose methylprednisolone given once a month during the washout period for the switch between natalizumab and fingolimod, compared to that of a placebo, on multiple sclerosis inflammatory rebound evaluated using MRI, 16 to 18 weeks after natalizumab discontinuation and clinically at 6 months

SECONDARY OUTCOMES:
comparison of the number of new T2 or gadolinium enhanced lesions on MRI in the 2 treatment groups | at 4 months
comparison of the number of MS relapses during the 6 months after natalizumab discontinuation, in the 2 treatment groups | at 6 months
potential correlations between previous MS activity and the risk of relapse or inflammatory rebound on MRI after natalizumab discontinuation | at 6 months
  To study the potential correlations between previous MS activity (annualised relapse rate during the year before natalizumab initiation) and the risk of relapse or inflammatory rebound on MRI after natalizumab discontinuation, in the whole group
adverse effects of high dose oral prednisolone | at 6 months
use of methylprednisolone once every 4 weeks during the switch between natalizumab and fingolimod in patients with MS | at 6 months
  To perform a cost utility analysis in order to evaluate the use of methylprednisolone once every 4 weeks during the switch between natalizumab and fingolimod in patients with MS

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVELOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France